CLINICAL TRIAL: NCT06429280
Title: Clinical Data Registry of Amblyopia Patients on Luminopia Treatment
Status: Recruiting | Type: Observational
Sponsor: Luminopia (Industry)
Responsible Party: Sponsor
Other Study IDs: R-AM-1
Record Dates: First submitted 2024-02-23; First posted 2024-05-24 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: N/A this is an observational study of Standard of Care — Medical Device which treats unilateral amblyopia through therapeutic software which stimulate vision

SUMMARY:
Amblyopia is the most prevalent cause of reduced monocular visual acuity in children and young adults, with estimates of prevalence ranging from 1% to 5%. The most common associated amblyogenic risk factors are uncorrected anisometropia, strabismus, or a combination of these. In addition to reduced visual acuity, amblyopic patients may also have measurable dysfunction of accommodation, fixation, binocularity, vergence, reading fluency, depth perception, and contrast sensitivity.

For the first time since the incorporation of atropine penalization into amblyopia management, physicians can now offer Luminopia, an FDA-approved dual action dichoptic treatment, to patients with amblyopia. Since the product became commercially available in November 2022, the number of patients on Luminopia therapy continues to grow. This presents a unique opportunity to gather real world evidence from a large number of patients, representative of how ophthalmologists and optometrists are applying this novel treatment in the real world. A registry of the clinical data associated with Luminopia treatment, with IRB oversight, will provide answers to key scientific questions using a large dataset.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of amblyopia
* Have undergone or currently undergoing Luminopia treatment for a minimum of 12 weeks

Exclusion Criteria:

-Have participated in prior Luminopia clinical trials

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a diagnosis of Amblyopia
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Acuity from baseline to consecutive visits | 3, 6,12, 24 months
  Change in Visual Acuity from baseline to consecutive visits
Duration of Visual Acuity treatment and number of follow-up visits | 3, 6,12, 24 months
  Duration of Visual Acuity treatment and number of follow-up visits
Durability of Visual Acuity results post-treatment cessation | 3, 6,12, 24 months
  Durability of Visual Acuity results post-treatment cessation
Adherence with Luminopia treatment | 3, 6,12, 24 months
  Adherence with Luminopia treatment
Change in Stereoacuity from baseline to consecutive visits | 3, 6,12, 24 months
  Change in Stereoacuity from baseline to consecutive visits

SECONDARY OUTCOMES:
Visual Acuity analyses will also be conducted by Prior Treatment | 3, 6,12, 24 months
  Visual Acuity analyses will also be conducted by Prior Treatment
Visual Acuity analyses will also be conducted by Amblyopia Type | 3, 6,12, 24 months
  Visual Acuity analyses will also be conducted by Amblyopia Type
Visual Acuity Analyses will also be conducted by Age | 3, 6,12, 24 months
  Visual Acuity Analyses will also be conducted by Age
Visual Acuity analyses will also be conducted by Baseline Angle of Deviation | 3, 6,12, 24 months
  Visual Acuity analyses will also be conducted by Baseline Angle of Deviation
Visual Acuity analyses will also be conducted by Severity (Baseline Visual Acuity) | 3, 6,12, 24 months
  Visual Acuity analyses will also be conducted by Severity (Baseline Visual Acuity)
Visual Acuity analyses will also be conducted by Adherence to Treatment | 3, 6,12, 24 months
  Visual Acuity analyses will also be conducted by Adherence to Treatment
Visual Acuity Analyses will also be conducted by Prescribed Dose | 3, 6,12, 24 months
  Visual Acuity Analyses will also be conducted by Prescribed Dose

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - UCSF Benioff Children's Physicians, San Ramon, California
  - Sansum Clinic, Santa Barbara, California
  - Okaloosa Ophthalmology, Crestview, Florida
  - Family Focus Eye Care, Gainsville, Florida
  - Eye Physicians of Central Florida, Maitland, Florida
  - Children's Eye Institute of Savannah, Savannah, Georgia
  - Honolulu Eye Clinic, Honolulu, Hawaii
  - Lurie Children's Hospital, Chicago, Illinois
  - Riley Children's Hospital at IU Health, Indianapolis, Indiana
  - Nevada Eye Physicians, Las Vegas, Nevada
  - Concord Eye Center, Concord, New Hampshire
  - Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - Pediatric Eye Specialist, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No